CLINICAL TRIAL: NCT05784584
Title: A Prospective, Observational, Cohort, Multicenter Study of Early Anti-Retroviral Treatment in HIV- Infected Infants
Brief Title: Early Anti-Retroviral Treatment in HIV- Infected Children
Status: Completed | Type: Observational
Sponsor: PENTA Foundation (Network)
Responsible Party: Sponsor
Other Study IDs: EARTH
Record Dates: First submitted 2023-03-02; First posted 2023-03-27 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: HIV Infections
Keywords: HIV; Infection; Infants; Antiretroviral Therapy
MeSH Terms: conditions — HIV Infections; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Infants infected through breast-feeding and perinatally: Infants infected through breast-feeding and perinatally diagnosed with HIV ≤90 days of age and starting ART ≤90 days after diagnosis. For these patients clinical data and blood for viral load, immunology and serology will be collected in the 11 visits.
  Interventions: Procedure: Blood samples collection

INTERVENTIONS:
Procedure: Blood samples collection — The study population will take blood samples for virological and immunological measurements.

SUMMARY:
EARTH study is conducted as part of the EPIICAL project. It is a prospective cohort study which aims to monitor clinical, virological and immunological features of HIV-positive, early treated children (≤90 days after diagnosis), in order to identify participants with excellent viral and immunological control, and also other without excellent control, in order to stratify potential participants in proof-of-concept trials directed to HIV cure.

DETAILED DESCRIPTION:
The duration of the study is 4 years from the start of enrollment with at least 4 years of follow-up for each participant. The study is conducted in South Africa, Mali, and Mozambique with an expected enrollment target of 200 participants (as a minimum). In this study, newly diagnosed HIV-infected children will start ART as early as possible, following local standards of care, and will be followed up to 4 years of age. Clinical and blood data for viral load, immunology, and serology will be collected at the 11 visits. HIV reservoir size and HIV-specific immune responses will be analyzed at visit 1 and at 1, 2, 3, and 4 years after enrollment. We will identify children with HIV infection eligible to participate in proof-of-concept treatment/remission studies.

A predictive model developed from European participant data will help identify children with low reservoir. These predictions will then be compared with available data from participants already enrolled with an excellent control to refine the model.

ELIGIBILITY:
Inclusion Criteria:

1. Perinatally infected infants who start ART at ≤90 days after diagnosis (HIV infection diagnosed and confirmed by molecular methods in 2 different samples, i.e., positive qualitative HIV DNA/RNA test).
2. Breastfed-infected children found to be infected ≤ 90 days of age and who started ART at < 90 days after diagnosis. This group will be younger than six months of age at ART initiation.
3. Caregivers (mother, if alive and available) able to provide informed consent.
4. Able to take ART.

Exclusion Criteria:

1. Second and successive RNA PCR negative
2. Malignancy
3. Current concomitant immunosuppressive therapy (including>15 days and >2 mg/kg/day of prednisone-equivalent).
4. Caregivers withdraw consent
5. Age >180 days.

Max Age: 180 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Perinatally infected infants who begin ART ≤ 90 days after diagnosis. Breastfed infants diagnosed with HIV ≤90 days of age and starting ART ≤ 90 days after diagnosis.
  The diagnosis of HIV transmission by breastmilk will be made from infants who:
  1. Have a negative birth HIV PCR
  2. Are being breastfed
  3. Who subsequently have 2 molecular methods positive for HIV. These tests will be conducted selectively among participants with a clinical evaluation suggestive of HIV infection, at the discretion of the attending physician.
Sampling Method: Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-03-28 (Actual)

PRIMARY OUTCOMES:
Proportion of children with excellent HIV control | 4 years
  Proportion of children with excellent HIV control profile at 2 and 4 years of age. This excellent control profile includes a composite endpoint of all of the following:
  1. Undetectable HIV RNA viral load in peripheral blood in the last year (blips, spikes and suboptimal viral control allowed, see below for definitions),
  2. Reservoir size (Total DNA /million PBMC) below 25th percentile with ddPCR / IPDA.
  3. Good immunological control (defined as a CD4 >30% and a good NK or CTL response) during the last year

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Tagarro, MD, Study Chair — Fundación Investigación Hospital 12 de Octubre
Locations (6):
- Centre Hospitalier Universitaire Gabriel Touré, Bamako, Mali
- Mozambique (2):
  - Centro de Investigaçao em Saude de Manhiça, Manica
  - Fundação Ariel Glaser contra o SIDA Pediátrico, Maputo
- South Africa (3):
  - Tygerberg Children's Hospital (TCH), Cape Town
  - Africa Health Research Institute (AHRI), Durban
  - PHRU, Soweto

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-21): https://cdn.clinicaltrials.gov/large-docs/84/NCT05784584/Prot_SAP_000.pdf